Optimized Camera-based Patient Positioning in CT: Impact on Radiation Exposure.

ClinicalTrials.gov ID: NCT05135208 29-August-2022

## **Study Protocol and Statistical Analysis Plan**

Title: Optimized Camera-based Patient Positioning in CT: Impact on Radiation Exposure.

Description of the study:

To investigate different options for patient positioning. Target parameters are the achievable differences in radiation exposure and the deviation from isocenter.

Design:

Retrospective

Status: The patients are positioned laser guided on the CT table by the trained technicians for the CT examinations.

A 128-slice single-source CT scanner was used. This CT scanner system with an integrated 3D camera system offers a recommendation for the patient's table positioning.

Statistical analysis

For radiation exposure analysis:

Power analysis was performed with a sample size of 1806 patients for each group to detect an effective size of 0.12 for radiation exposure analysis based on test measurements on an anthropomorphic phantom.

Isocenter accuracy:

According to previous results, a power analysis for the isocenter accuracy was performed with a group size of 10 patients in each group.

A chi-squared test was used to analyze patients' characteristics.

Levine's test was used for calculating the equality of variances followed by student's t-test for independent samples. A p value < 0.05 was considered indicating statistically significant differences. For the study, the patients are not additionally exposed to radiation or contrast media. Tests that require a higher radiation exposure (perfusion) are excluded.

The evaluation of the data is carried out anonymously via a dose management system.

The duration of the study will be approximately 12 months.

## Results:

| | Cameramode | Н | Mean value | Standard- deviation | P valu |
|---|---|---|---|---|---|
| isocenter | off | 1557 | -10.9 | 16.6 | 0.000 |
| | on | 1561 | -3.8 | 10.1 | |
| Reconstruction diameter | off | 1557 | 400.8 | 40.8 | 0.251 |
| | on | 1561 | 399.2 | 40.1 | |
| pitch | off | 1557 | 0.8 | 0.2 | 0.894 |
| | on | 1561 | 0.8 | 0.2 | |
| mAS max | off | 1557 | 219.8 | 114.2 | 0.042 |
| | on | 1561 | 211.2 | 112.2 | |
| kVp | off | 1557 | 94.8 | 18.6 | 0.796 |
| | on | 1561 | 95.0 | 18.8 | |
| Table height | off | 1557 | 170.0 | 20.4 | 0.000 |
| | on | 1561 | 165.6 | 16.2 | |
| age | off | 1557 | 64.1 | 15.8 | 0.423 |
| | on | 1561 | 63.7 | 16.1 | |
| вмі | off | 1557 | 26.1 | 5.4 | 0.957 |
| | on | 1561 | 26.1 | 5.5 | |
| weight | off | 1557 | 76.2 | 18.4 | 0.885 |
| | on | 1561 | 76.3 | 18.0 | |
| height | off | 1557 | 1704.6 | 97.8 | 0.506 |
| | on | 1561 | 1707.0 | 96.4 | |

## Legend:

mAs = milliampere-seconds; kVp = kilovoltage peak; BMI= Body Mass Index

| | Cameramode | Н | Mean value | Standard-<br>deviation | P value |
|---|---|---|---|---|---|
| ED | off | 1557 | 3.5 | 2.9 | 0.053 |
| | on | 1561 | 3.3 | 2.7 | |
| DLP | off | 1557 | 342.0 | 280.7 | 0.033 |
| | on | 1561 | 321.1 | 266.7 | |
| CTDI <sub>vol</sub> | off | 1557 | 6.8 | 4.6 | 0.011 |
| | on | 1561 | 6.4 | 4.3 | |
| Organ dose of eye lens | off | 1557 | 0.1 | 0.1 | 0.21 |
| | on | 1561 | 0.1 | 0.3 | |
| Organ dose of<br>heart | off | 1557 | 3.9 | 3.1 | 0.443 |
| | on | 1561 | 3.8 | 3.0 | |
| Organ dose of colon | off | 1557 | 3.5 | 3.9 | 0.015 |
| | on | 1561 | 3.1 | 3.6 | |
| Organ dose of ovaries | off | 1557 | 3.1 | 3.6 | 0.902 |
| | on | 1561 | 3.1 | 3.5 | |
| Organ dose of red bone marrow | off | 1557 | 2.4 | 2.1 | 0.049 |
| | on | 1561 | 2.3 | 1.9 | |
| Organ dose of thyroid gland | off | 1557 | 0.3 | 0.4 | 0.305 |
| | on | 1561 | 0.3 | 0.8 | 0.205 |
| Organ dose of upper colon | off | 1557 | 3.7 | 3.9 | 0.012 |
| | on | 1561 | 3.3 | 3.6 | |
| Organ dose of salivary glands | off | 1557 | 0.0 | 0.0 | 0.226 |
| | on | 1561 | 0.0 | 0.2 | |
| Organ dose of esophagus | off | 1557 | 2.3 | 1.7 | 0.355 |
| | on | 1561 | 2.2 | 1.7 | |

Legends: Dose Length Product (DLP) in mGy\*cm, Effective Dose (ED) in mSv, CT Dose Index  $(CTDI_{vol}) \ in \ mGy_{\overline{\tau}} \ and \ Organ \ Dose \ in \ mSv.$